CLINICAL TRIAL: NCT06954948
Title: Effect of a Home-Based Pulmonary Rehabilitation on Patients' Outcome With COPD In Limited Recourses Country
Brief Title: Effect of Home-Based Pulmonary Rehabilitation
Acronym: PR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Newroz Ghazi Aziz, Assist Professor, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: home-based PR
Record Dates: First submitted 2025-04-10; First posted 2025-05-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: COPD
Keywords: COPD; Exacerbation; 6MWD; CAT; mMRC; CRQ; Pulmonary Rehabilitation; MARS-5
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Pre-post test will be adopted to assess the difference in the clinical outcomes of 64 staple patients with COPD after home-based pulmonary rehabilitation compared with 64 patients in control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COPD (Experimental): 64 stable COPD patients receive eight week structured pulmonary rehabilitation program. Two session per week (1-2 hours) with continuous phon call. participants will be given structured manual. Primary outcomes are changes in the exacerbation rate, functional status and mMRC. Secondary outcomes are improvement in the health related quality of life and medication adherence with correct use of inhaler. To validate internal consistency all the outcomes will be compared with 64 patients in control group.
  Interventions: Behavioral: pulmonary rehabilitation (PR)

INTERVENTIONS:
Behavioral: pulmonary rehabilitation (PR) — PR is an exercise and education programme designed for people with lung disease who experience symptoms of breathlessness.

SUMMARY:
This clinical trial aims to assess the effectiveness of home-based pulmonary rehabilitation in improving the clinical outcomes of patients with COPD.

Research questions :

RQ1: Is there a significant difference in the exacerbation rates before and after implementing the program? RQ2: Is there a significant improvement in the quality of life before and after implementing the program? RQ3: Is there a significant improvement in 6MWT before and after implementing the program? RQ4: Is there a significant improvement in COPD patients' modified Medical Research Council dyspnea scale before and after the implementation of the program?

Intervention group will receive pulmonary rehabilitation at home or any place they designated over eight consecutive weeks. Two sessions per week and continuous phone calls. Participants will also be given a structured manual to record their activities and follow instructions on days without supervision. While the control group receive routine care at the respiratory unit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD, confirmed by spirometry and pulmonologist
* Age ≥40 years (to avoid recruiting participants with asthma rather than COPD)
* Current or previous smoker (≥10 packs per year)
* Confidence in using the proposed pulmonary rehabilitation (PR) system
* Kurdish language fluency
* Willingness to participate and sign an informed consent form.

Exclusion Criteria:

* patients with pulmonary hypertension
* patients with movement disorders and/or a history of falls
* patients with severe sensory or cognitive impairment
* patients with symptomatic ischemic heart disease
* patients with musculoskeletal degenerative disease
* Patients out site of the city or inability to be contacted

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Exacerbation rate | eight weeks after the implementation of the program
  A COPD exacerbation, or flare-up, occurs when COPD respiratory symptoms become much more severe.
Functional status (exercise capacity) | eight weeks after the program implementation
  The functional status is measured by the mean difference in the six minute walking distance (6MWD)
mMRC | eight weeks after the program implementation
  modified Medical Research Council (mMRC) dyspnea scale is self-reported tool used to assess the severity of breathlessness and it's effect on the activity of daily living when the COPD patients is in the stable condition. The score of 0 demonstrates that the patient has the lowest breathlessness and no restriction to activities and the score of 4 shows that the patient has severe breathlessness and greatest impairment.

SECONDARY OUTCOMES:
CAT | eight weeks after the program implementation
  The COPD Assessment Test™ (CAT) is a self-reported questionnaire that helps patients and healthcare professional to measure the impact that COPD (Chronic Obstructive Pulmonary Disease) is having on patients' wellbeing and daily life. The CAT score is the total of the scores from the eight assessed areas. The maximum score is 40 and it is categorized based on the severity as the follows.
  0-9 low impact 0-20 medium impact 21-30 high impact 31-40 very high impact
Chronic Respiratory Questionnaire (CRQ) | eight weeks after the program implementation
  The CRQ is a disease-specific health-related quality of life questionnaire, developed to measure the impact of Chronic Obstructive Pulmonary Disease (COPD) on a person's life. This tool is self-completed questionnaire, it has 20 items, 4 domains (Dyspnea, Fatigue, Emotional Function & Mastery). The scaling of items is 7-pointing modified Likert Scale (1-7) and 0-7 on dyspnea domain. Higher score indicates better quality of life.
Medication adherence assessment with MARS-5 | eight weeks after the program implementation
  The MARS-5 Item Questionnaire The MARS-5 questionnaire consists of five questions on forgetting, changing dosage, stopping, skipping, and taking less medication. The score ranges from 5 to 25, where a higher MARS-5 score indicates higher self-reported adherence. One item assesses unintentional non-adherence and four items assess intentional non-adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University, Erbil, Kurdistan, Iraq

IPD SHARING:
Plan to Share IPD: No